CLINICAL TRIAL: NCT06170840
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of QY101 Ointment in Patients With Plaque Psoriasis
Brief Title: A Study of QY101 Ointment in Subjects With Plaque Psoriasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: E-nitiate Biopharmaceuticals (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QY101-Ⅱ-1
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- QY101 placebo ointment (Placebo Comparator): 40 subjects use QY101 placebo ointment twice daily for 12 weeks
  Interventions: Drug: QY101Placebo/QY101 ointment
- 0.3% QY101 ointment (Experimental): 60 subjects use QY101 placebo ointment twice daily for 12 weeks
  Interventions: Drug: QY101Placebo/QY101 ointment
- 1.0 % QY101 ointment (Experimental): 60 subjects use1.0 % QY101 ointment twice daily for 12 weeks
  Interventions: Drug: QY101Placebo/QY101 ointment

INTERVENTIONS:
Drug: QY101Placebo/QY101 ointment — External use for BID

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of QY101 ointment in adult patients with plaque psoriasis (2-20% BSA).

DETAILED DESCRIPTION:
Participants will be stratified and randomly assigned to trial groups two (Test group 1:0.3%; Test group 2:1.0%, 60 patients per group) or placebo group (40 patients) according to the ratio of 3:3:2 and BSA (BSA < 10% or BSA ≥ 10%) . All groups will be receive with QY101 ointment or placebo, treatment for twice daily (BID) for 12 weeks; All subjects are required to take part in visit at 2, 4, 6, 8 and 12 weeks, they were followed up for efficacy assessment, safety examination and pharmacokinetics samples collection (with week 8 as the primary efficacy endpoint), and safety follow-up was administered 28 ± 7 days after the last dose via telephone .

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and comply with the test process, voluntarily participate in the test and provide informed consent;
2. When signing the informed consent, age ≤ 18 years old ≤ 75 years old, gender is not limited;
3. The patient meets the diagnosis of plaque psoriasis, has a history of plaque psoriasis for ≥ 6 months before randomization, and meets the following conditions:

   1. At baseline, plaque psoriasis covered 2% to 20% of BSA (including both ends) (scalp, palms, and soles were not counted as BSA);
   2. Physician overall assessment (PGA) ≥ 2 at baseline;
4. Fertile men and women of childbearing age must agree to use reliable contraception from the time they sign an informed consent until six months after the last dose of the investigational drug; Blood pregnancy tests for women of childbearing age must be negative during screening and at baseline.

Exclusion Criteria:

1. Other types of psoriasis were diagnosed during screening, such as gutting psoriasis, erythrodermic psoriasis, generalized pustular psoriasis, arthropathic psoriasis, drug-induced or drug-aggravated psoriasis;
2. The presence of other systemic autoimmune inflammatory diseases and skin lesions (such as eczema), which may affect the evaluation of treatment outcomes;
3. Subjects who are expected to receive additional local therapy, phototherapy, or other systemic therapy other than investigational medication during the trial;
4. Taking drugs that can aggravate psoriasis (such as lithium, antimalarial drugs, etc.);
5. Patients who have failed or are intolerant to previous treatment with Phosphodiesterase-4 (PDE4) inhibitors;
6. Known to be allergic to the study drug or related excipients (QY101 ointment and excipients: albuvarin, light liquid paraffin, propylene glycol, Carbonic acid, glyceryl behenate, glyceryl monodistearate, hydroxyphenyl butyl, propyl gallate and disodium edetate), or have a history of angioedema or allergy to topical drugs;
7. receive contraindicated drugs, supplements, and other treatments prescribed in this trial that may affect the course of psoriasis within the specified time period prior to initial dosing or planned for the duration of the trial (see Appendix 2: Concomitant medications during the trial);
8. Participants who are participating in another interventional clinical trial or whose last use of another investigational drug is less than 5 half-lives prior to the first dosing of the investigational drug;
9. any history of infection or recurrent infection requiring systemic antibiotic treatment within 2 weeks prior to first dosing, or serious infection requiring hospitalization or intravenous antibiotic treatment within 8 weeks prior to first dosing (e.g., pneumonia, cellulitis, bone or joint infection, etc.); Recurrent, chronic, or other active infection at the time of initial dosing, if the investigator determines that participation in the study increases participants' risk;
10. Use of a suppressant of CYP3A liver metabolic enzyme, or use of any medication, including prescription, over-the-counter, and herbal oral or topical drugs, other than vitamins and/or Paracetamol, within 2 weeks prior to initial administration;
11. Participants who have received, or plan to receive, a live or attenuated vaccine within 4 weeks prior to initial administration;
12. Abnormal laboratory test results during screening, including:

    1. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or basic phosphoric acid

       Enzyme (ALP) > 2.5 × Upper Limit of Normal (ULN);
    2. Serum creatinine > 1.5×ULN, or creatinine clearance < 50 mL/min.
13. Hepatitis B surface antigen (HBsAg) positive or hepatitis B core antibody (HBcAb) positive, and hepatitis B virus deoxyribonucleic acid (HBV-DNA) positive; Or hepatitis C virus (HCV) antibody positive and HCV-RNA positive; Or positive for HIV, Treponema Pallidum-Antibody (TP-Ab) (Rapid Plasma Reagin, TP-AB) RPR] or Toluidine Red Unheated Serum Test (except for negative Toluidine Red Unheated Serum Test, TRUST);
14. The presence of decompensated cardiac insufficiency (New York Heart Disease Assocation (NYHA) class III or IV) within 6 months prior to screening; History of unstable angina pectoris, myocardial infarction, coronary artery bypass grafting or coronary stent implantation; There are severe arrhythmias that require medication or cardiac assistance, such as degree II type 2 or degree III atrioventricular block, long QT Interval, or long QT block. QT syndrome or Fridericia Corrected QT Interval (QTcF) abnormality (male > 470 ms female > 480 ms) corrected according to the Fridericia formula and assessed by the investigator as unsuitable for participation in this clinical trial; Hospitalization due to Cardiovascular (CV) events, CV disease or CV surgery; Peripheral artery disease diagnosed by angiography with stroke (ischemic or hemorrhagic, including transient ischemic attack) should be excluded;
15. Known malignant tumors or history of malignant tumors (excluding clinically cured skin basal cell carcinoma, skin squamous cell carcinoma, cervical carcinoma in situ);
16. Patients with psychoneuro-related diseases or history (such as depression, epilepsy), which affect medication compliance or the researcher's clinical judgment of suicide risk;
17. Pregnant or lactating women, female subjects or male subjects' partners planning to become pregnant (within 6 months after signing the informed consent to the last administration of the study drug);
18. Other conditions deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Physician Global Assessment（PGA）response | 8 weeks
  At week 8, the proportion of subjects in each trial group who responded to the Physician Global Assessment (PGA) compared to the placebo group.
  The PGA response was defined as a PGA score of 0 (clear) or 1 (nearly clear) and an improvement of ≥ 2 points from baseline on the PGA scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided